CLINICAL TRIAL: NCT00674414
Title: A Phase II, Randomized, Multi-center Study, Assessing Value of Adding Everolimus (RAD001) to Trastuzumab as Preoperative Therapy of HER-2 Positive Primary Breast Cancer Amenable to Surgery.
Brief Title: Trastuzumab With or Without Everolimus in Treating Women With Breast Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IDMC decision due to accrual issue (82 pts accrued / 120 expected)
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595159; FRE-FNCLCC-GEP-04/0606-RAD-HER; EUDRACT-2007-004098-24; EU-20851
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Everolimus

ARMS (2):
- Arm I (Active Comparator): Patients receive trastuzumab (Herceptin®) IV once weekly for 6 weeks. Patients then undergo surgery.
  Interventions: Biological: trastuzumab; Procedure: therapeutic conventional surgery
- Arm II (Experimental): Patients receive trastuzumab as in arm I and oral everolimus once daily for 6 weeks. Within 24 hours after completing everolimus, patients undergo surgery.
  Interventions: Biological: trastuzumab; Drug: everolimus; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: trastuzumab — Trastuzumab (Herceptin®) IV once weekly
Drug: everolimus — Oral everolimus once daily
  Arms: Arm II
Procedure: therapeutic conventional surgery — Patients undergo surgery

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether giving everolimus together with trastuzumab is more effective than giving trastuzumab alone in treating women with breast cancer.

PURPOSE: This randomized phase II trial is studying trastuzumab and everolimus to see how well they work compared to trastuzumab alone before surgery in treating patients with breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the added efficacy obtained by the association of trastuzumab (Herceptin®) with everolimus as preoperative therapy of primary HER2-positive breast cancer as shown by increased clinical tumor response rate.

Secondary

* To compare the inhibition of the two pathways, RAS/RAF/MAP kinase and PI3-kinase/AKT/mTor.
* To evaluate whether the pre-treatment molecular characteristics of tumor and serum or their modifications early in the treatment are predictive of clinical response.
* To compare the frequency of pathological complete response achieved in the two groups after 6 weeks of treatment.
* To determine disease-free survival at 3 years.
* To evaluate safety and tolerability of the two treatment regimens.
* To analyze the possible relationships between treatment toxicity and constitutional gene polymorphisms linked to the administered agents.
* To analyze the possible relationships between response and molecular pharmacodynamic assessments, including proteomics (blood samples), Bio-Plex protein array (tumor), and IHC (tumor).
* To analyze the drug levels and pharmacokinetic assessments of everolimus and trastuzumab (Herceptin®).

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive trastuzumab (Herceptin®) IV once weekly for 6 weeks. Patients then undergo surgery.
* Arm II: Patients receive trastuzumab as in arm I and oral everolimus once daily for 6 weeks. Within 24 hours after completing everolimus, patients undergo surgery.

Blood and tumor samples are collected periodically during study for pharmacogenomic, proteomic, and pharmacokinetic studies.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of invasive breast cancer

  * Previously untreated disease
* Candidate for breast-conserving surgery, as defined by both of the following:

  * Clinical stage cT1-3, cN0-2 disease
  * Clinical stage M0 disease (bone scan, chest X-ray, and liver ultrasound required at screening to exclude metastatic disease)
* HER2-positive primary tumor, defined as meeting either of the following criteria:

  * IHC 3+
  * IHC 2+ and FISH positive (centralized confirmation)
* No inflammatory breast cancer or bilateral breast cancer

  * Patients who have been treated for cancer of the contralateral breast can be included if there is at least a 5 year time interval from last systemic treatment for breast cancer before randomization into this study
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Menopausal status not specified
* WBC ≥ 3.5 x 10^9/L
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hb ≥ 10 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum transaminases activity ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* FEV > 55% by MUGA or ECHO
* Spirometry and DLCO > 50% of normal
* O_2 saturation > 88% at rest on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to everolimus, sirolimus, trastuzumab (Herceptin®), or lactulose
* No hypercholesterolemia/hypertriglyceridemia ≥ grade 3

  * No hypercholesterolemia/hypertriglyceridemia ≥ grade 2 with history of coronary artery disease (despite lipid-lowering treatment if given)
* No uncontrolled infection
* No other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including any of the following:

  * Uncontrolled hypertension
  * Congestive cardiac failure
  * Ventricular arrhythmias
  * Active ischemic heart disease
  * Myocardial infarction within the past year
  * Chronic liver or renal disease
  * Active gastrointestinal tract ulceration
  * Severely impaired lung function
* No known history of HIV seropositivity
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Willing to participate in the biological investigations
* Not deprived of liberty or placed under guardianship
* Patients must be affiliated to a Social Security System

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days (from the screening visit) since prior other investigational drugs
* More than 5 days (from randomization) since prior and no concurrent strong inhibitors or inducers of the isoenzyme CYP3A, including any of the following

  * Rifabutin
  * Rifampicin
  * Clarithromycin
  * Ketoconazole
  * Itraconazole
  * Voriconazole
  * Ritonavir
  * Telithromycin
* No other concurrent anti-cancer treatments such as chemotherapy, immunotherapy/biological response modifiers, endocrine therapy, or radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by clinical and echographic tumor evaluation | january 2013

SECONDARY OUTCOMES:
Disease-free survival at 3 years | January 2015
Pathological response assessed after 6 weeks of treatment | January 2013
Clinical response predictive factors | May 2013
Rate of pathological complete response (pCR) | January 2013
Pharmacogenomics, proteomics, immunohistochemistry (IHC), pharmacokinetics | december 2013
Toxicity as assessed by the standard NCI CTC-AE v3.0 scale | January 2013

CONTACTS AND LOCATIONS:
Overall Officials: Mario Campone, MD, Principal Investigator — Centre Regional Rene Gauducheau
Locations (8):
- France (8):
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Campone M, Bachelot T, Treilleux I, Pistilli B, Salleron J, Seegers V, Arnedos M, Loussouarn D, Wang Q, Vanlemmens L, Jimenez M, Rios M, Dieras V, Leroux A, Paintaud G, Rezai K, Andre F, Lion M, Merlin JL. A phase II randomised study of preoperative trastuzumab alone or combined with everolimus in patients with early HER2-positive breast cancer and predictive biomarkers (RADHER trial). Eur J Cancer. 2021 Nov;158:169-180. doi: 10.1016/j.ejca.2021.09.017. Epub 2021 Oct 19. PMID 34678678